CLINICAL TRIAL: NCT00055601
Title: A Phase II Randomized Trial for Patients With Muscle-Invading Bladder Cancer Evaluating Transurethral Surgery and BID Irradiation Plus Either Paclitaxel and Cisplatin or 5-Fluorouracil and Cisplatin Followed by Selective Bladder Preservation and Gemcitabine/Paclitaxel/Cisplatin Adjuvant Chemotherapy
Brief Title: Combination Chemotherapy and Radiation Therapy With/Without Surgery In Patients With Stage II/III Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0233; CDR0000258303; ECOG-R0233; NCI-2011-01578 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Fluorouracil; Paclitaxel; Radiotherapy; Gemcitabine; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic RT + paclitaxel + cisplatin (Experimental): Induction: Twice-daily pelvic radiation therapy (RT) with paclitaxel and cisplatin; Consolidation: Twice-daily pelvic radiation therapy with paclitaxel and cisplatin if tumor response is T0/Ta/Tis or radical cystectomy if tumor response is ≥ T1; Adjuvant: gemcitabine, paclitaxel, and cisplatin.
  Interventions: Drug: cisplatin; Drug: paclitaxel; Radiation: radiation therapy; Drug: Gemcitabine; Procedure: Radical cystectomy
- Pelvic RT + fluorouracil + cisplatin (Experimental): Induction: Twice-daily pelvic radiation therapy (RT) with fluoruracil and cisplatin; Consolidation: Twice-daily pelvic radiation therapy with fluoruracil and cisplatin if tumor response is T0/Ta/Tis or radical cystectomy if tumor response is ≥ T1; Adjuvant: gemcitabine, paclitaxel, and cisplatin.
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy; Drug: Gemcitabine; Procedure: Radical cystectomy

INTERVENTIONS:
Drug: cisplatin — Induction: 15 mg/m2 as a 60-minute infusion on days 1, 2, 3, 8, 9, 10, 15, 16, and 17; Consolidation: 15 mg/m2 as a 60-minute infusion on days 1, 2, 8, and 9; Adjuvant: 35 mg/m2 as a 60-minute infusion on days 1 and 8 of each 21-day cycle for 4 cycles.
Drug: fluorouracil — Induction: 400 mg/m2 as a 24-hour infusion on days 1, 2, 3, 15, 16, and 17; Consolidation: 400 mg/m2 as a 24-hour infusion on days 1, 2, 3, 8, 9, and 10.
  Arms: Pelvic RT + fluorouracil + cisplatin
Drug: paclitaxel — Induction: 50 mg/m2 as a 60-minute infusion on days 1, 8, and 15; Consolidation: 50 mg/m2 as a 60-minute infusion on days 1 and 8; Adjuvant: 50 mg/m2 as a 60-minute infusion on days 1 and 8 of each 21-day cycle for 4 cycles.
  Arms: Pelvic RT + paclitaxel + cisplatin
Radiation: radiation therapy — Induction: External beam irradiation, 1.6 Gy, will be given to the pelvis in the first treatment followed by an interfraction period of at least 4-6 hours. During the second treatment, 1.5 Gy will be delivered to the whole bladder for the first five sessions (7.5 Gy) then to the tumor plus a margin for eight sessions (12. Gy). Consolidation: Consolidation therapy will start 7-14 days following a cystoscopic re-evaluation demonstrating a complete response to the induction therapy. 1.5 Gy (per fraction) will be given to the pelvis in two treatment fractions per day, with an interfraction period of at least 4-6 hours.
Drug: Gemcitabine — Adjuvant: 1000 mg/m2 over 30-60 minutes on days 1 and 8 of each 21-day cycle for 4 cycles.
Procedure: Radical cystectomy — Operable patients with pT1 or worse tumor response on re-evaluation following induction therapy will have radical cystectomy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy (RT) uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of combination chemotherapy plus radiation therapy with or without surgery is more effective in treating bladder cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of two combination chemotherapy regimens and radiation therapy with or without radical cystectomy in treating patients who have stage II or stage III bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the safety and tolerability of induction paclitaxel, cisplatin, and radiotherapy or fluorouracil, cisplatin, and radiotherapy followed by consolidation chemoradiotherapy or radical cystectomy and adjuvant gemcitabine, paclitaxel, and cisplatin in patients with operable stage II or III bladder cancer.
* Estimate the efficacy of these regimens, in terms of complete response, in patients who have undergone prior transurethral resection (TUR).
* Estimate the efficacy of these regimens after TUR, in terms of preserving the native tumor-free bladder 5 years after therapy, in these patients.
* Estimate the function of the preserved bladder in patients treated with these regimens after TUR.
* Determine the value of tumor histopathologic, molecular genetic, and DNA content parameters as possible prognostic factors for initial tumor response and recurrence-free survival in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to T stage (T2 vs T3/T4 ). Patients are randomized to one of two treatment arms.

* Induction therapy (weeks 1-3):

  * Arm I: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and cisplatin IV over 1 hour on days 1-3, 8-10, and 15-17. Patients also receive pelvic radiotherapy twice daily on days 1-5, 8-12, and 15-17.
  * Arm II: Patients receive fluorouracil IV over 24 hours on days 1-3 and 15-17 and cisplatin IV over 1 hour on days 1-3, 8-10, and 15-17. Patients also receive pelvic radiotherapy as in arm I.

Patients in both arms who achieve complete response after induction therapy proceed to consolidation therapy on week 8. Patients with operable pT1 or worse tumor response proceed to radical cystectomy on week 9.

* Consolidation therapy (weeks 8 and 9):

  * Arm I: Patients receive paclitaxel IV over 1 hour on days 1 and 8 and cisplatin IV over 1 hour on days 1, 2, 8, and 9. Patients also receive pelvic radiotherapy twice daily on days 1-5 and 8-10.
  * Arm II: Patients receive 5-FU IV over 24 hours on days 1-3 and 8-10 and cisplatin as in arm I. Patients also receive radiotherapy as in arm I.
* Adjuvant chemotherapy (weeks 21-33 or 17-29): Beginning 12 weeks after consolidation therapy or 8 weeks after radical cystectomy, patients receive gemcitabine IV over 30-60 minutes, paclitaxel IV over 1 hour, and cisplatin IV over 1 hour on days 1 and 8. Treatment repeats every 3 weeks for 4 courses.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 96 patients (48 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed operable primary muscle invasive bladder cancer

  * T2-T4a, NX or N0, M0 (stage II or III)
* Must have an adequate functioning bladder
* Must have undergone a prior transurethral resection of the bladder tumor within the past 8 weeks
* No evidence of tumor-related hydronephrosis
* No evidence of distant metastases or histologically or cytologically confirmed lymph node metastases
* Patients with involvement of the prostatic urethra with transitional cell cancer that was visibly completely resected are allowed

  * No evidence of stromal invasion of the prostate

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin at least 10 g/dL
* White blood cell (WBC) count at least 4,000/mm^3
* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Serum bilirubin no greater than 2.0 mg/dL

Renal

* Serum creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min NOTE: If the creatinine clearance is greater than 60 mL/min, creatinine of no greater than 1.8 mg/dL is allowed at the discretion of the study chair

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer, stage T1a prostate cancer, or carcinoma in situ of the cervix
* Must be able to tolerate systemic chemotherapy with pelvic radiotherapy and radical cystectomy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* See Disease Characteristics

Other

* No concurrent drugs that have potential nephrotoxicity or ototoxicity (e.g., aminoglycosides)

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-12 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L. Zietman, MD, Principal Investigator — Massachusetts General Hospital; Robert Uzzo, MD, Study Chair — Fox Chase Cancer Center; Robert Dreicer, MD, FACP, Study Chair — The Cleveland Clinic
Locations (2):
- United States (2):
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Mak RH, Hunt D, Shipley WU, Efstathiou JA, Tester WJ, Hagan MP, Kaufman DS, Heney NM, Zietman AL. Long-term outcomes in patients with muscle-invasive bladder cancer after selective bladder-preserving combined-modality therapy: a pooled analysis of Radiation Therapy Oncology Group protocols 8802, 8903, 9506, 9706, 9906, and 0233. J Clin Oncol. 2014 Dec 1;32(34):3801-9. doi: 10.1200/JCO.2014.57.5548. Epub 2014 Nov 3. PMID 25366678
- [Derived] Mitin T, Hunt D, Shipley WU, Kaufman DS, Uzzo R, Wu CL, Buyyounouski MK, Sandler H, Zietman AL. Transurethral surgery and twice-daily radiation plus paclitaxel-cisplatin or fluorouracil-cisplatin with selective bladder preservation and adjuvant chemotherapy for patients with muscle invasive bladder cancer (RTOG 0233): a randomised multicentre phase 2 trial. Lancet Oncol. 2013 Aug;14(9):863-72. doi: 10.1016/S1470-2045(13)70255-9. Epub 2013 Jul 1. PMID 23823157

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic RT + Paclitaxel + Cisplatin: Induction: Twice-daily pelvic radiation therapy with paclitaxel and cisplatin; Consolidation: Twice-daily pelvic radiation therapy with paclitaxel and cisplatin if tumor response is T0/Ta/Tis or radical cystectomy if tumor response is ≥ T1; Adjuvant: gemcitabine, paclitaxel, and cisplatin IV.
- Pelvic RT + Fluorouracil + Cisplatin: Induction: Twice-daily pelvic radiation therapy with fluoruracil and cisplatin; Consolidation: Twice-daily pelvic radiation therapy with fluoruracil and cisplatin if tumor response is T0/Ta/Tis or radical cystectomy if tumor response is ≥ T1; Adjuvant: gemcitabine, paclitaxel, and cisplatin IV.
Period: Overall Study
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin
Started | 48 | 49
Completed | 46 (Subjects with data available for the primary analysis are considered to have completed the study.) | 47 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — No protocol treatment received | 1 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients who started protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 82] | 67 [44 to 83] | 66 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion Rate
Description: Radiation therapy and chemotherapy per protocol or within acceptable variation guidelines based on central review. The study was designed for a two-sided binomial test with 87% power and a significance level of 0.05 with a null hypothesis of a 70% completion rate against the alternative 90% completion rate. For each arm, more than 34 out of 43 evaluable patients completing the treatment, would indicate to reject the null hypothesis for a better treatment completion rate. Fewer than 24 out 43 evaluable patients completing the treatment would indicate to reject the null hypothesis for a worse treatment completion rate. Otherwise, the conclusion would be that there is not enough evidence to reject the null hypothesis of a 70% completion rate in either direction.
Time Frame: From randomization to 11 weeks
Population: All eligible patients who started study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin
Number analyzed (Participants) | 46 | 47
percentage of participants | 67 [51 to 80] | 53 [38 to 68]

2. Secondary Outcome: Complete Response After Induction
Description: Complete response requires the absence of any tumor in the tumor-site biopsy specimen or elsewhere and a bimanual exam that does not indicate the presence of a tumor mass.
Time Frame: From randomization to eight weeks
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin
Number analyzed (Participants) | 46 | 47
percentage of participants | 72 [57 to 84] | 62 [46 to 76]

3. Secondary Outcome: Bladder-intact Survival Rate (5 Years)
Description: Bladder-intact survival was measured from the date of randomization to occurrence of cystectomy or death. Five-year rates were estimated using the Kaplan-Meier method.
Time Frame: From the date of randomization to five years.
Population: All eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin
Number analyzed (Participants) | 46 | 47
percentage of participants | 67 [53 to 81] | 71 [57 to 84]

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. the same methodology was applied for non-serious adverse events (AE).
Arm/Group | Pelvic RT + Paclitaxel + Cisplatin | Pelvic RT + Fluorouracil + Cisplatin
Serious Adverse Events (participants affected / at risk) | 43/46 | 39/47
Other Adverse Events (participants affected / at risk) | 46/46 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pelvic RT + Paclitaxel + Cisplatin (N=46) | Pelvic RT + Fluorouracil + Cisplatin (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Hematologic-Other (Blood and lymphatic system disorders) | 3 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 | 3
Hemoglobin for leukemia (Blood and lymphatic system disorders) | 0 | 1
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 6 | 6
Platelet transfusion (Blood and lymphatic system disorders) | 0 | 1
Circulatory or cardiac-Other (Cardiac disorders) | 0 | 1
Edema NOS (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Ventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Constitutional symptons-Other (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pain-other (General disorders) | 1 | 0
Culture wound positive (Infections and infestations) | 0 | 2
Infection NOS (Infections and infestations) | 1 | 4
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 | 2
Infection with unknown ANC (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Leukopenia NOS (Investigations) | 8 | 10
Lymphopenia (Investigations) | 4 | 10
Neutropenia (Investigations) | 27 | 18
Neutrophils/granulocytes for leukemia (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 16 | 11
Weight increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Blood magnesium decreased (Metabolism and nutrition disorders) | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 8 | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Ataxia NEC (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (exc vertigo) (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Anxiety NEC (Psychiatric disorders) | 1 | 0
Depression NEC (Psychiatric disorders) | 1 | 0
Bladder disorder NOS (Renal and urinary disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 1
Hematuria present (Renal and urinary disorders) | 2 | 1
Late RT toxicity: Bladder: NOS (Renal and urinary disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 1 | 1
Renal/GU-Other (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 3
Urinary frequency (Renal and urinary disorders) | 2 | 4
Urinary incontinence (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Pelvic pain NOS (Reproductive system and breast disorders) | 0 | 1
Urogenital fistula (Reproductive system and breast disorders) | 0 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin-Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hemorrhage NOS (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis NOS (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pelvic RT + Paclitaxel + Cisplatin (N=46) | Pelvic RT + Fluorouracil + Cisplatin (N=47)
Hematologic-Other (Blood and lymphatic system disorders) | 26 | 19
Hemoglobin decreased (Blood and lymphatic system disorders) | 43 | 43
Hemolysis NOS (Blood and lymphatic system disorders) | 3 | 1
Circulatory or cardiac-Other (Cardiac disorders) | 4 | 1
Edema NOS (Cardiac disorders) | 7 | 7
Palpitations (Cardiac disorders) | 1 | 3
Hearing impaired (Ear and labyrinth disorders) | 4 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 18 | 22
Diarrhea (with colostomy) (Gastrointestinal disorders) | 1 | 3
Diarrhea NOS (Gastrointestinal disorders) | 33 | 36
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Flatulence (Gastrointestinal disorders) | 3 | 1
GI-other (Gastrointestinal disorders) | 9 | 4
Late RT toxicity: Bowel: NOS (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 27 | 28
Proctalgia (Gastrointestinal disorders) | 1 | 3
Proctitis NOS (Gastrointestinal disorders) | 2 | 4
Rectal bleeding (Gastrointestinal disorders) | 6 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 6
Vomiting NOS (Gastrointestinal disorders) | 7 | 16
Chest pain (General disorders) | 1 | 3
Constitutional symptons-Other (General disorders) | 1 | 3
Fatigue (General disorders) | 41 | 44
Injection site reaction NOS (General disorders) | 2 | 3
Late RT toxicity: Other: NOS (General disorders) | 12 | 8
Pain-other (General disorders) | 10 | 11
Pyrexia (General disorders) | 6 | 4
Rigors (General disorders) | 3 | 5
Hepatic-Other (Hepatobiliary disorders) | 5 | 6
Infection NOS (Infections and infestations) | 2 | 5
Alanine aminotransferase increased (Investigations) | 12 | 10
Aspartate aminotransferase increased (Investigations) | 10 | 10
Blood alkaline phosphatase NOS increased (Investigations) | 8 | 9
Blood bilirubin increased (Investigations) | 7 | 6
Blood creatinine increased (Investigations) | 21 | 17
Leukopenia NOS (Investigations) | 41 | 37
Lymphopenia (Investigations) | 8 | 8
Metabolic-Other (Investigations) | 12 | 5
Neutropenia (Investigations) | 16 | 18
Platelet count decreased (Investigations) | 30 | 33
Weight decreased (Investigations) | 4 | 5
Weight increased (Investigations) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 18 | 19
Blood albumin decreased (Metabolism and nutrition disorders) | 9 | 12
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 5 | 3
Blood magnesium decreased (Metabolism and nutrition disorders) | 22 | 17
Dehydration (Metabolism and nutrition disorders) | 14 | 8
Hyperglycemia NOS (Metabolism and nutrition disorders) | 19 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 9
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 13
Hypokalemia (Metabolism and nutrition disorders) | 4 | 7
Hyponatremia (Metabolism and nutrition disorders) | 16 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Dizziness (exc vertigo) (Nervous system disorders) | 13 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 13 | 6
Taste disturbance (Nervous system disorders) | 8 | 7
Anxiety NEC (Psychiatric disorders) | 7 | 4
Insomnia NEC (Psychiatric disorders) | 16 | 11
Dysuria (Renal and urinary disorders) | 15 | 11
Hematuria present (Renal and urinary disorders) | 5 | 7
Late RT toxicity: Bladder: NOS (Renal and urinary disorders) | 17 | 17
Renal/GU-Other (Renal and urinary disorders) | 11 | 12
Urinary frequency (Renal and urinary disorders) | 29 | 31
Urinary retention (Renal and urinary disorders) | 4 | 1
Impotence (Reproductive system and breast disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 10
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 5 | 5
Skin-Other (Skin and subcutaneous tissue disorders) | 3 | 1
Flushing (Vascular disorders) | 4 | 1
Hypotension NOS (Vascular disorders) | 2 | 3
Phlebitis superficial (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.